CLINICAL TRIAL: NCT00178659
Title: Proteomics of Brain Trauma-associated Elevated Intracranial Pressure (ICP)
Acronym: Proteomics
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: TIRR/Mission Connect (Other); The Center for Clinical and Translational Sciences (CCTS) Clinical Research Unit at The University of Texas Health Science Center at Houston (Other)
Responsible Party: Principal Investigator, Georgene Hergenroeder, Associate Professor, Neurosurgery, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-04-040; N-13-04-040
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Brain Injuries, Traumatic; Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI (Traumatic Brain Injury); Proteomics
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples for use in identifying proteins related to head trauma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1 healthy volunteers: Healthy volunteers to act as controls - Recruitment is complete for this cohort
  Interventions: Other: Blood/saliva samples for protein/molecular analysis
- 2 head trauma: Head trauma patients meeting enrollment criteria - Recruitment is complete for this cohort
  Interventions: Other: Blood/saliva samples for protein/molecular analysis
- 3 orthopedic injury: The orthopedic injury cohort will include patients admitted to the ED able to provide informed consent with the following:
  1. Fracture confirmed radiographically
  2. No head trauma
  3. No other known inflammatory process or infection
  4. No history of neurological or psychiatric disorders or alcohol or drug dependency
  Interventions: Other: Blood/saliva samples for protein/molecular analysis
- 4 Mild TBI: The mild TBI patients will be defined as those admitted to the ED experiencing, - Recruitment is complete for this cohort
  1. Non-penetrating head trauma manifesting one or more of the following:
     * Loss of consciousness
     * Post-traumatic amnesia
     * Altered mental status
     * Focal neurologic deficits, seizure
  2. GCS> 12
  3. No abnormalities on CT other than contusion
  4. No operative Lesions
  5. Length of hospital stay < 48 hrs
  6. No other known inflammatory process or infection
  7. No history of neurological or psychiatric disorders or alcohol or drug dependency
  Interventions: Other: Blood/saliva samples for protein/molecular analysis

INTERVENTIONS:
Other: Blood/saliva samples for protein/molecular analysis — Bloods samples - healthy volunteers(1 time) head injury subjects (5 times). Blood and/or saliva samples mild TBI patients (2 times) and healthy volunteers (2 times)
  Other Names: blood samples; saliva samples

SUMMARY:
The specific aim of this research is to determine if the blood from brain-injured patients contains reproducible protein markers that appear prior to elevations in intracranial pressure (ICP).

DETAILED DESCRIPTION:
One of the major causes of death following brain trauma is increased intracranial pressure (ICP). Currently, there are no effective ways to predict if the ICP of a patient will reach uncontrollable levels. Various cytokines (balance between pro-and anti-inflammatory) and other factors are thought to underlie increases in ICP. The specific aim of this research is to determine if the blood from brain-injured patients contains reproducible protein markers that appear prior to elevations in ICP. We propose to employ mass spectrometry, antibody array and ELISA to profile proteins in the serum of patients suffering from traumatic brain injury. These protein profiles will be compiled by a pattern recognition program that has the capacity to learn and make predictions based on the spectra and associated patient information. Each time a sample is analyzed, it is added to the database allowing the program to make increasingly accurate predictions. Protein profiles of patients with known ICP values will be analyzed. Our hypothesis is that alterations in serum protein composition will precede changes in intracranial pressure giving rise to predictable patterns that can be detected using large-scale proteomic analysis. After approximately 90 non-brain trauma and 90 brain-trauma patients are analyzed, if markers are found, the predictability of elevated ICP will be tested. If successful, this may aid the neurosurgeon in determining future courses of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 14-65 years old
* Non-penetrating brain injury
* ICP monitor or
* Healthy volunteer or

The orthopedic injury cohort will include patients admitted to the ED able to provide informed consent with the following:

1. Fracture confirmed radiographically
2. No head trauma
3. No other known inflammatory process or infection
4. No history of neurological or psychiatric disorders or alcohol or drug dependency.

or The mild TBI patients will be defined as those experiencing,

1. Non-penetrating head trauma manifesting one or more of the following:

   * Loss of consciousness
   * Post-traumatic amnesia
   * Altered mental status
   * Focal neurologic deficits, seizure
2. GCS> 12
3. No abnormalities on CT other than contusion
4. No operative Lesions
5. Length of hospital stay < 48 hrs
6. No other known inflammatory process or infection
7. No history of neurological or psychiatric disorders or alcohol or drug dependency

Exclusion Criteria:

* Inability to obtain informed consent

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consenting healthy volunteers, head trauma, mild head trauma or acute orthopedic injury patients meeting enrollment criteria listed below.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Elevated intracranial pressure | within the first 10 days post injury
  Intracranial pressure >20mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Dash, PhD, Principal Investigator — The University of Texas, Houston
Locations (1):
- The University of Texas, Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available

REFERENCES:
- [Background] Redell JB, Moore AN, Ward NH 3rd, Hergenroeder GW, Dash PK. Human traumatic brain injury alters plasma microRNA levels. J Neurotrauma. 2010 Dec;27(12):2147-56. doi: 10.1089/neu.2010.1481. Epub 2010 Nov 23. PMID 20883153
- [Background] Hergenroeder GW, Moore AN, McCoy JP Jr, Samsel L, Ward NH 3rd, Clifton GL, Dash PK. Serum IL-6: a candidate biomarker for intracranial pressure elevation following isolated traumatic brain injury. J Neuroinflammation. 2010 Mar 11;7:19. doi: 10.1186/1742-2094-7-19. PMID 20222971
- [Background] Hergenroeder G, Redell JB, Moore AN, Dubinsky WP, Funk RT, Crommett J, Clifton GL, Levine R, Valadka A, Dash PK. Identification of serum biomarkers in brain-injured adults: potential for predicting elevated intracranial pressure. J Neurotrauma. 2008 Feb;25(2):79-93. doi: 10.1089/neu.2007.0386. PMID 18260791